CLINICAL TRIAL: NCT01700699
Title: Impact of BRAFV600E Intratumor Heterogeneity on the Efficacy of Tyrosine Kinase Inhibitors in the Treatment of Radioiodine-resistant Thyroid Cancer
Brief Title: Impact of BRAFV600E Intratumor Heterogeneity in Thyroid Cancer Treated With Tyrosine Kinase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Mario Vitale, Professor of Endocrinology at the School of Medicine, University of Salerno, Director of the Endocrinology Unit, University Hospital of Salerno, Italy, University of Salerno
Other Study IDs: BRAF-TKI-DTC1
Record Dates: First submitted 2012-09-22; First posted 2012-10-04 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Differentiated Thyroid Cancer
Keywords: thyroid cancer; tyrosine kinase inhibitors; BRAF; Sorafenib; Pazopanib; Sunitinib; Cabozantinib
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Primary and metastatic tumor tissue, frozen or formaldehyde fixed-paraffin embedded from block, genomic DNA already extracted from tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Sorafenib: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with Sorafenib
- Axitinib: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with Axitinib
- Pazopanib: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with Pazopanib
- TKI: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with different type of tyrosine kinase inhibitor
- Motesanib: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with Motesanib
- Sunitinib: Assessment of percentage of BRAFV600E in tissue specimens of MRR-DTC patients treated with Sunitinib

SUMMARY:
* Background: BRAFV600E is the most frequent oncogene in differentiated thyroid cancer (DTC) occurring in about 50% of cases. Clinical trials with tyrosine kinase inhibitors (TKI) with specific activity against BRAF in metastatic radioiodine-resistant DTC (MRR-DTC) are ongoing. Very recently it has been demonstrated that DTC often consists of a mixture of tumor cells with wild-type and mutant BRAF. The subclonal occurrence of BRAFV600E in MRR-DTC could disable the therapy with BRAF targeted TKI and be responsible of the frequent defeats of this treatment. A therapeutic strategy based upon BRAF inhibitors in tumors bearing subclonal BRAFV600E could be initially successful hitting the tumor cells expressing the oncogene, and after the initial tumor growth arrest and/or shrinkage, the oncogene negative cells insensitive or less sensitive to the treatment, could restart the growth of the tumor causing the progression of the disease and the escape from the clinical response.
* Aims: To determine the impact of subclonal BRAFV600E on the efficacy of BRAF inhibitors in the treatment of MRR-DTC.
* Study design: Primary tumor tissues will be analyzed for the presence of BRAFV600E by pyrosequencing or other quantitative assay. If available, synchronous metastases and post-therapy metachronous metastases will be analyzed as well. The clinical response will be determined according to RECIST, and the association with the percentage of BRAFV600E alleles will be evaluated. Attention will be paid to the possible difference of BRAFwild-type/BRAFV600E ratio between primary tumors and synchronous metastases, primary tumors and post-therapy metachronous metastases, and between responsive and resistant synchronous tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

* subjects any sex any age with metastatic or unresectable thyroid carcinoma treated with tyrosine kinase inhibitors
* evidence of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
* availability of study end points including best response, duration of response, and time to disease progression (based on RECIST), clinical progression, or death
* availability of tumor tissue samples, frozen or formaldehyde fixed-paraffin embedded from block, genomic DNA already extracted from tumor tissue

Exclusion Criteria:

* concurrent Hashimoto's thyroiditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of BRAFV600E alleles in tumor tissue before TKI treatment | within 1 month after the patient has entered the study

SECONDARY OUTCOMES:
Percentage of BRAFV600E alleles in tumor tissue post-TKI treatment | within 30 days from the availability of the tissue sample

CONTACTS AND LOCATIONS:
Overall Officials: Mario Vitale, MD, Principal Investigator — Univeristy of Salerno, Italy
Locations (1):
- Department of Medicine and Surgery, Univeristy of Salerno, Baronissi, Salerno, Italy

REFERENCES:
- [Background] Guerra A, Fugazzola L, Marotta V, Cirillo M, Rossi S, Cirello V, Forno I, Moccia T, Budillon A, Vitale M. A high percentage of BRAFV600E alleles in papillary thyroid carcinoma predicts a poorer outcome. J Clin Endocrinol Metab. 2012 Jul;97(7):2333-40. doi: 10.1210/jc.2011-3106. Epub 2012 Apr 16. PMID 22508706
- [Background] Guerra A, Sapio MR, Marotta V, Campanile E, Rossi S, Forno I, Fugazzola L, Budillon A, Moccia T, Fenzi G, Vitale M. The primary occurrence of BRAF(V600E) is a rare clonal event in papillary thyroid carcinoma. J Clin Endocrinol Metab. 2012 Feb;97(2):517-24. doi: 10.1210/jc.2011-0618. Epub 2011 Dec 14. PMID 22170714
- [Background] Gupta-Abramson V, Troxel AB, Nellore A, Puttaswamy K, Redlinger M, Ransone K, Mandel SJ, Flaherty KT, Loevner LA, O'Dwyer PJ, Brose MS. Phase II trial of sorafenib in advanced thyroid cancer. J Clin Oncol. 2008 Oct 10;26(29):4714-9. doi: 10.1200/JCO.2008.16.3279. Epub 2008 Jun 9. PMID 18541894
- [Background] Kloos RT, Ringel MD, Knopp MV, Hall NC, King M, Stevens R, Liang J, Wakely PE Jr, Vasko VV, Saji M, Rittenberry J, Wei L, Arbogast D, Collamore M, Wright JJ, Grever M, Shah MH. Phase II trial of sorafenib in metastatic thyroid cancer. J Clin Oncol. 2009 Apr 1;27(10):1675-84. doi: 10.1200/JCO.2008.18.2717. Epub 2009 Mar 2. PMID 19255327